CLINICAL TRIAL: NCT01940471
Title: A Phase 3, Randomized, Double-Blind Study to Evaluate the Safety and Efficacy of Tenofovir Alafenamide (TAF) 25 mg QD Versus Tenofovir Disoproxil Fumarate (TDF) 300 mg QD for the Treatment of HBeAg-Positive, Chronic Hepatitis B
Brief Title: Study to Compare Tenofovir Alafenamide (TAF) Versus Tenofovir Disoproxil Fumarate (TDF) in Participants With Chronic Hepatitis B Infection Who Are Positive for Hepatitis B e Antigen
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-320-0110; 2013-000636-10 (EudraCT Number)
Record Dates: First submitted 2013-08-20; First posted 2013-09-12 (Estimated); Results first posted 2017-03-30 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-09

CONDITIONS: HBeAg-positive Chronic Hepatitis B
Keywords: Hepatitis; Tenofovir; Viread
MeSH Terms: conditions — Hepatitis | interventions — tenofovir alafenamide; Tenofovir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- TAF 25 mg (Experimental): TAF + TDF placebo for 96 weeks (per amendment 1 & 2) or 144 weeks (per amendment 3).
  Interventions: Drug: TAF; Drug: TDF Placebo
- TDF 300 mg (Active Comparator): TDF + TAF placebo for 96 weeks (per amendment 1 & 2) or 144 weeks (per amendment 3).
  Interventions: Drug: TDF; Drug: TAF Placebo
- Open-label TAF (Experimental): All participants who complete the double-blind period (96 weeks or 144 weeks) will be eligible to receive open-label TAF until Week 384 of the study.
  After the end of study treatment, participants can either switch to commercially available anti-HBV treatments in their country or will be followed every 4 weeks, for up to 24 weeks off treatment (treatment-free follow-up (TFFU)) for safety assessment.
  Interventions: Drug: TAF

INTERVENTIONS:
Drug: TAF — 25 mg tablet administered orally once daily
  Other Names: Vemlidy®; GS-7340
  Arms: Open-label TAF; TAF 25 mg
Drug: TDF — 300 mg tablet administered orally once daily
  Other Names: Viread®
  Arms: TDF 300 mg
Drug: TAF Placebo — Tablet administered orally once daily
  Arms: TDF 300 mg
Drug: TDF Placebo — Tablet administered orally once daily
  Arms: TAF 25 mg

SUMMARY:
The primary objective of this study is to compare the efficacy, safety, and tolerability of tenofovir alafenamide (TAF) versus tenofovir disoproxil fumarate (TDF) in treatment-naive and treatment-experienced adults with hepatitis B e antigen (HBeAg)-positive chronic hepatitis B virus (HBV) infection.

DETAILED DESCRIPTION:
This study GS-US-320-0110 is a multi-center clinical trial planned to enroll participants in multiple countries, including China. However, due to the review timeline difference in China, full enrollment was reached in the main study before China was able to participate. Therefore, details for the China cohort are registered separately (NCT02836249) on ClinicalTrials.gov as this cohort will not be part of the main study analysis.

ELIGIBILITY:
Key Inclusion Criteria:

* Ability to understand and sign a written informed consent form, which must be obtained prior to initiation of study procedures.
* Adult males and non-pregnant, non-lactating females.
* Documented evidence of chronic HBV infection.
* HBeAg-positive, chronic hepatitis B with all of the following:

  * HBeAg-positive at screening.
  * Screening HBV DNA ≥ 2 x 10^4 IU/mL
  * Screening serum alanine aminotransferase (ALT) level > 60 U/L (males) or > 38 U/L (females) and ≤ 10 x the upper limit of the normal range (ULN).
* Treatment-naive participants (defined as < 12 weeks of oral antiviral treatment with any nucleoside or nucleotide analogue) OR treatment-experienced participants (defined as participants meeting all entry criteria [including HBV DNA and serum ALT criteria] and with ≥ 12 weeks of previous treatment with any nucleoside or nucleotide analogue).
* Previous treatment with interferon (pegylated or non-pegylated) must have ended at least 6 months prior to the baseline visit.
* Adequate renal function.
* Normal electrocardiogram (ECG).

Key Exclusion Criteria:

* Females who are breastfeeding.
* Males and females of reproductive potential who are unwilling to use an "effective", protocol specified method(s) of contraception during the study.
* Co-infection with hepatitis C virus, human immunodeficiency virus (HIV), or hepatitis D virus.
* Evidence of hepatocellular carcinoma .
* Any history of, or current evidence of, clinical hepatic decompensation.
* Abnormal hematological and biochemical parameters, including aspartate aminotransferase (AST) > 10 x ULN.
* Received solid organ or bone marrow transplant.
* History of malignancy within the past 5 years, with the exception of specific cancers that are cured by surgical resection; individuals under evaluation for possible malignancy are not eligible.
* Currently receiving therapy with immunomodulators (eg, corticosteroids), investigational agents, nephrotoxic agents, or agents capable of modifying renal excretion.
* Individuals receiving ongoing therapy with drugs not to be used with tenofovir alafenamide or tenofovir disoproxil fumarate or individuals with a known hypersensitivity to study drugs, metabolites, or formulation excipients.
* Current alcohol or substance abuse judged by the investigator to potentially interfere with participant compliance.
* Any other clinical condition or prior therapy that, in the opinion of the Investigator, would make the participant unsuitable for the study or unable to comply with dosing requirements.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 875 (Actual)
Dates: Start 2013-09-11 (Actual); Primary Completion 2015-11-16 (Actual); Study Completion 2022-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (159):
- United States (15):
  - Coalition of Inclusive Medicine, Los Angeles, California
  - Stanford University Medical Center, Palo Alto, California
  - Huntington Medical Research Institutes, Pasadena, California
  - Research and Education, Inc., San Diego, California
  - Silicon Valley Research Institute, San Jose, California
  - University of Miami, Miami, Florida
  - Digestive Disease Associates, PA, Catonsville, Maryland
  - Tufts Medical Center, Inc, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Sing Chan Private Practice, Flushing, New York
  - New Discovery, LLC, Flushing, New York
  - Jefferson Medical College, Philadelphia, Pennsylvania
  - Xiaoli Ma, PC, Philadelphia, Pennsylvania
  - Texas Clinical Research Institute, LLC, Arlington, Texas
  - Kelsey Research Foundation, Houston, Texas
- Australia (11):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Westmead Hospital Westmead, Westmead, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Monash Medical Centre, Clayton, Victoria
  - St. Vincent's Hospital, Fitzroy, Victoria
  - Footscray Hospital, Footscray, Victoria
  - Austin Health, Heidelberg, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- Bulgaria (4):
  - Tokuda Hospital - Sofia, Sofia
  - MHAT Alexandrovska Medical University, Sofia, Sofia
  - MMA Hospital of Active Treatment, Sofia
  - MHAT Sofia Med, Sofia
- Canada (12):
  - University of Calgary, Calgary, Alberta
  - Zeidler Ledcor Centre Division of Gastroenterology / Department of Medicine, Edmonton, Alberta
  - Liver and Intestinal Research Centre, Vancouver, British Columbia
  - Gordon and Leslie Diamond Health Care Centre, Vancouver, British Columbia
  - Dr. John Farley, Inc., Vancouver, British Columbia
  - Vancouver Infectious Disease Research and Care Centre, Vancouver, British Columbia
  - Gastrointestinal Research Institute (GIRI), Vancouver, British Columbia
  - University of Manitoba, Health Sciences Center, Winnipeg, Manitoba
  - The Ottawa Hospital, Ottawa, Ontario
  - University Health Network / Toronto General Hospital, Toronto, Ontario
  - Inspiration Research Limited, Toronto, Ontario
  - Toronto Liver Centre, Toronto, Ontario
- France (4):
  - Hopital Beaujon, Clichy
  - Hopital Pitie Salpetriere, Paris
  - Hopital Civil de Strasbourg, Strasbourg
  - Hopital Paul Brousse, Villejuif
- Hong Kong (5):
  - Queen Mary Hospital, Hong Kong
  - Princess Margaret Hospital, Lai Chi Kok
  - Prince of Wales Hospital, Shatin
  - Alice Ho Miu Ling Nethersole Hospital, Tai Po
  - Tuen Mun Hospital, Tuenmen
- India (18):
  - BYL Nair Hospital & T N Medical College, Mumbai, Maharashtra
  - Government Medical College and Superspecialty Hospital, Nagpur, Maharashtra
  - Midas Multispecialty Hospital, Nagpur, Maharashtra
  - SMS Medical College & Hospital, Jaipur, Rajasthan
  - Postgraduate Institute of Medical Education & Research, Chandigarh
  - YR Gaitonde Centre for AIDS Research and Education, Chennai
  - VGM Hospital, Coimbatore
  - Gleneagles Global Hospital, Hyderabad
  - Centre for Liver Research & Diagnostic, Deccan College of Medical Sciences and Allied Hospitals, Hyderabad
  - S. R Kalla Memorial Gastro & General Hospital, Jaipur
  - Peerless Hospital & B.K.Roy Research Center, Kolkata
  - Postgraduate Institute of Medical Education & Research, Kolkata
  - Seth GS Medical College and KEM Hospital, Mumbai
  - All India Institute of Medical Sciences, New Delhi
  - Sir Ganga Ram Hospital, New Delhi
  - Institute of Liver and Biliary Sciences, New Delhi
  - Global Hospital Super Specialty & Transplant Centre, Pārel
  - Nirmal Hospital, Surat
- Italy (7):
  - Azienda Ospedaliera di Bologna - Policlinico S. Orsola Malpighi, Bologna
  - Istituto Europeo di Oncologia, Bologna
  - Azienda Ospedaliero Universitaria Ospedali Riuniti di, Foggia
  - Policlinico Universitario G. Martino via Consolare, Messina
  - Azienda Ospedale San Paolo, Milan
  - Azienda Ospedaliera di Padova, Padua
  - Azienda Ospedaliero Universitaria Pisana, Pisa
- Japan (16):
  - Kyushu University Hospital, Fukuoka, Fukuoka-shi
  - Shin-Kokura Hospital, Fukuoka
  - National Hospital Organization Kyushu Medical Center, Fukuoka
  - Kagawa Prefectural Central Hospital, Kagawa
  - Kobe City Medical Center General Hospital, Kobe
  - Yamanashi Prefectural Central Hospital, Kofu
  - Kurume University Hospital, Kurume
  - Kyoto Prefectural University of Medicine, Kyoto
  - Japan Red Cross Musashino Hospital, Musashino
  - Hyogo College of Medicine, Nishinomiya
  - Okayama University Hospital, Okayama
  - Osaka Red Cross Hospital, Osaka
  - Osaka University Hospital, Osaka
  - National Hospital Organization Nagasaki Medical Center, Ōmura
  - Hokkaido University Hospital, Sapporo
  - Medical Hospital of Tokyo Medical and Dental University, Tokyo
- New Zealand (2):
  - Auckland Clinical Studies Limited, Auckland
  - Waikato Hospital (District Health Board), Hamilton
- Poland (5):
  - Uniwersytecki Szpital Kliniczny w Bialymstoku Klinika, Bialystok
  - Szpital Specjalistyczny, Chorzów
  - SPZOZ, Wojewódzki Specjalistyczny Szpital, Lodz
  - SP ZOZ Wojewódzki Szpital Zakazny, Warsaw
  - Centrum Badan Klinicznych, Wroclaw
- Romania (5):
  - Institutul National de Boli Infectioase "Prof. Dr. Matei Bals", Bucharest
  - Centrul Medical de Diagnostic si Tratament "Dr. Victor Babes", Bucharest
  - Spitatul Clinic de Boli Infectioase Constanta, Constanța
  - Gastromedica SRL, Iași
  - Spitalul Clinic Judetean de Urgenta Timisoara, Timișoara
- Russia (11):
  - Lipetsk Regional Center for Prevention and Control of AIDS and Infectious Diseases, Lipetsk
  - Scientific Research Institute of Nutrition, Moscow
  - People's Friendship University of Russia, Moscow
  - 1st Moscow State Medical University University Clinical Hospital #3, Moscow
  - Limited Liability Company "Modern Medicine Clinic", Moscow
  - Institute of Clinical Immunology RAMS, Clinic of Immunopathology, Novosibirsk
  - Scientific Research Institute of Clinical Immunology, Novosibirsk
  - Municipal Clinical Hospital n.a. S.P. Botkin, Saint Petersburg
  - Research Institute of Influenza, Saint Petersburg
  - Medical Company Hepatology, Samara
  - Sverdlovsk Regional Clinical Hospital #1, Yekaterinburg
- Singapore (3):
  - National University Hospital Singapore, Singapore
  - Singapore General Hospital, Singapore
  - Changi General Hospital Pte Ltd., Singapore
- South Korea (22):
  - Kosin University College of Medicine, Busan, Seo-gu
  - Pusan National University Hospital, Busan
  - SoonChunHyang University Hospital Cheonan, Cheonan
  - Keimyung University Dongsan Medical Center, Daegu
  - Kyungpook National University Hospital, Daegu
  - Konyang University Hospital, Daejeon
  - Inje University Ilsan Paik Hospital, Gyeonggi-do
  - Ajou University Hospital, Gyeonggi-do
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Seoul Saint Mary Hospital, Seoul
  - Asan Medical Center, Seoul
  - Konkuk University Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
  - Chung-Ang University Hospital, Seoul
  - Ulsan University Hospital, Ulsan
  - Yonsei Unversity Wonju, Wŏnju
  - Pusan National University Yangsan Hospital, Yangsan
- Spain (2):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Virgen del Rocio, Seville
- Taiwan (8):
  - Chiayi Christian Hospital, Chiayi City
  - Hualien Tzu Chi Medical Center, Hualien City
  - Kaohsiung Med. College Hosp. Dept. of Internal Medicine, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Cathay General Hospital, Taipei
  - Far-Eastern Memorial Hospital, Taipei
- Turkey (Türkiye) (5):
  - Ankara Üniversitesi Gastroenteroloji Bilim Dalı Cebeci, Ankara
  - University of Uludag, Bursa
  - Dicle University Medical Faculty Department of Infectious Diseases, Diyarbakır
  - Istanbul Universitesi Cerrahpassa Tip Fakultesi Enfeksiyon, Istanbul
  - Ege Universitesi Tip Fakultesi Hastanesi, Izmir
- United Kingdom (4):
  - Barts & The London NHS Trust, London
  - Royal Free Hospital, London
  - King's College Hospital, London
  - Nottingham University Hospitals NHS Trust, Nottingham

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gileadclinicaltrials.com/transparency-policy/
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gileadclinicaltrials.com/transparency-policy/

REFERENCES:
- [Derived] Buti M, Lim YS, Chan HLY, Agarwal K, Marcellin P, Brunetto MR, Chuang WL, Janssen HLA, Fung SK, Izumi N, Jablkowski MS, Abdurakhmanov D, Abramov F, Wang H, Botros I, Yee LJ, Mateo R, Flaherty JF, Osinusi A, Pan CQ, Shalimar X, Seto WK, Gane EJ. Eight-year efficacy and safety of tenofovir alafenamide for treatment of chronic hepatitis B virus infection: Final results from two randomised phase 3 trials. Aliment Pharmacol Ther. 2024 Dec;60(11-12):1573-1586. doi: 10.1111/apt.18278. Epub 2024 Sep 27. PMID 39327857
- [Derived] Lim YS, Chan HLY, Ahn SH, Seto WK, Ning Q, Agarwal K, Janssen HLA, Pan CQ, Chuang WL, Izumi N, Fung S, Shalimar, Brunetto M, Hui AJ, Chang TT, Lim SG, Abramov F, Flaherty JF, Wang H, Yee LJ, Kao JH, Gane E, Hou J, Buti M. Tenofovir alafenamide and tenofovir disoproxil fumarate reduce incidence of hepatocellular carcinoma in patients with chronic hepatitis B. JHEP Rep. 2023 Jul 13;5(10):100847. doi: 10.1016/j.jhepr.2023.100847. eCollection 2023 Oct. PMID 37771546
- [Derived] Chan HLY, Buti M, Lim YS, Agarwal K, Marcellin P, Brunetto M, Chuang WL, Janssen HLA, Fung S, Izumi N, Abdurakhmanov D, Jablkowski M, Celen MK, Ma X, Caruntu F, Flaherty JF, Abramov F, Wang H, Camus G, Osinusi A, Pan CQ, Shalimar, Seto WK, Gane E; GS-US-320-0110 and GS-US-320-0108 investigators. Long-Term Treatment With Tenofovir Alafenamide for Chronic Hepatitis B Results in High Rates of Viral Suppression and Favorable Renal and Bone Safety. Am J Gastroenterol. 2024 Mar 1;119(3):486-496. doi: 10.14309/ajg.0000000000002468. Epub 2023 Aug 9. PMID 37561058
- [Derived] Cathcart AL, Chan HL, Bhardwaj N, Liu Y, Marcellin P, Pan CQ, Shalimar, Buti M, Cox S, Parhy B, Zhou E, Martin R, Chang S, Lin L, Flaherty JF, Kitrinos KM, Gaggar A, Izumi N, Lim YS. No Resistance to Tenofovir Alafenamide Detected through 96 Weeks of Treatment in Patients with Chronic Hepatitis B Infection. Antimicrob Agents Chemother. 2018 Sep 24;62(10):e01064-18. doi: 10.1128/AAC.01064-18. Print 2018 Oct. PMID 30038044
- [Derived] Seto WK, Asahina Y, Brown TT, Peng CY, Stanciu C, Abdurakhmanov D, Tabak F, Nguyen TT, Chuang WL, Inokuma T, Ikeda F, Santantonio TA, Habersetzer F, Ramji A, Lau AH, Suri V, Flaherty JF, Wang H, Gaggar A, Subramanian GM, Mukewar S, Brunetto MR, Fung S, Chan HL. Improved Bone Safety of Tenofovir Alafenamide Compared to Tenofovir Disoproxil Fumarate Over 2 Years in Patients With Chronic HBV Infection. Clin Gastroenterol Hepatol. 2018 Jun 20:S1542-3565(18)30633-5. doi: 10.1016/j.cgh.2018.06.023. Online ahead of print. PMID 29933096
- [Derived] Agarwal K, Brunetto M, Seto WK, Lim YS, Fung S, Marcellin P, Ahn SH, Izumi N, Chuang WL, Bae H, Sharma M, Janssen HLA, Pan CQ, Celen MK, Furusyo N, Shalimar D, Yoon KT, Trinh H, Flaherty JF, Gaggar A, Lau AH, Cathcart AL, Lin L, Bhardwaj N, Suri V, Mani Subramanian G, Gane EJ, Buti M, Chan HLY; GS-US-320-0110; GS-US-320-0108 Investigators. 96 weeks treatment of tenofovir alafenamide vs. tenofovir disoproxil fumarate for hepatitis B virus infection. J Hepatol. 2018 Apr;68(4):672-681. doi: 10.1016/j.jhep.2017.11.039. Epub 2018 Jan 17. PMID 29756595
- [Derived] Chan HL, Fung S, Seto WK, Chuang WL, Chen CY, Kim HJ, Hui AJ, Janssen HL, Chowdhury A, Tsang TY, Mehta R, Gane E, Flaherty JF, Massetto B, Gaggar A, Kitrinos KM, Lin L, Subramanian GM, McHutchison JG, Lim YS, Acharya SK, Agarwal K; GS-US-320-0110 Investigators. Tenofovir alafenamide versus tenofovir disoproxil fumarate for the treatment of HBeAg-positive chronic hepatitis B virus infection: a randomised, double-blind, phase 3, non-inferiority trial. Lancet Gastroenterol Hepatol. 2016 Nov;1(3):185-195. doi: 10.1016/S2468-1253(16)30024-3. Epub 2016 Sep 22. PMID 28404091
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=GS-US-320-0110

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in East Asia, Europe, North America, Australia, India, and New Zealand.
Pre-assignment Details: 1396 participants were screened.
Groups:
- TAF 25 mg: Tenofovir alafenamide (Vemlidy®; TAF) 25 mg tablet + tenofovir disoproxil fumarate (Viread®; TDF) placebo tablet once daily for up to 96 weeks (per amendment 1 & 2) or 144 weeks (per amendment 3).
- TDF 300 mg: TDF 300 mg tablet + TAF placebo tablet once daily for up to 96 weeks (per amendment 1 & 2) or 144 weeks (per amendment 3).
- TAF 25 mg to TAF 25 mg: After Week 96 or 144 in the Blinded Treatment Phase, participants were given the option to continue with Open-label (OL) TAF 25 mg for additional 288 or 240 weeks (Up to Week 384), respectively.
  After the completion of OL TAF Extension Phase treatment or when there was early discontinuation of treatment, participants either switched to commercially available anti-HBV treatments in their country or entered follow-up phase and were followed-up every 4 weeks for 24 weeks off treatment (treatment-free follow-up [TFFU]) for the assessment of safety.
- TDF 300 mg to TAF 25 mg: After Week 96 or 144 in the Blinded Treatment Phase, participants were given the option to switch to OL TAF 25 mg for additional 288 or 240 weeks (Up to Week 384), respectively.
  After the completion of OL TAF Extension Phase treatment or when there was early discontinuation of treatment, participants either switched to commercially available anti-HBV treatments in their country or entered follow-up phase and were followed-up every 4 weeks for 24 weeks off treatment (TFFU) for the assessment of safety.
Period: Period 1: Double-blind Phase
Arm/Group | TAF 25 mg | TDF 300 mg | TAF 25 mg to TAF 25 mg | TDF 300 mg to TAF 25 mg
Started | 582 | 293 | 0 | 0
Completed | 515 | 253 | 0 | 0
Not Completed | 67 | 40 | 0 | 0
Not completed — Withdrew Consent | 31 | 18 | 0 | 0
Not completed — Lost to Follow-up | 8 | 6 | 0 | 0
Not completed — Investigator's Discretion | 8 | 5 | 0 | 0
Not completed — Pregnancy | 9 | 2 | 0 | 0
Not completed — Non-Compliance with Study Drug | 3 | 2 | 0 | 0
Not completed — Adverse Event | 2 | 2 | 0 | 0
Not completed — Death | 2 | 1 | 0 | 0
Not completed — Lack of Efficacy | 1 | 1 | 0 | 0
Not completed — Protocol-Specified Criteria for Withdrawal | 1 | 1 | 0 | 0
Not completed — Randomized but Never Treated | 1 | 1 | 0 | 0
Not completed — HbsAg Seroconversion | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Period: Period 2: Open-Label TAF Extension Phase
Arm/Group | TAF 25 mg | TDF 300 mg | TAF 25 mg to TAF 25 mg | TDF 300 mg to TAF 25 mg
Started (At the end of Double-blind Phase, participants were given the option to receive TAF in an OL TAF Extension Phase for up to 240 or 288 weeks.) | 0 | 0 | 514 (Out of 515 participants who completed the Double-blind Phase in TAF 25 mg arm, 1 participant did not enter the OL TAF Extension Phase.) | 253
Completed | 0 | 0 | 422 | 213
Not Completed | 0 | 0 | 92 | 40
Not completed — Withdrew Consent | 0 | 0 | 48 | 22
Not completed — Lost to Follow-up | 0 | 0 | 13 | 8
Not completed — Investigator's Discretion | 0 | 0 | 9 | 4
Not completed — Protocol-specified Criteria for Withdrawal | 0 | 0 | 5 | 4
Not completed — Adverse Event | 0 | 0 | 5 | 1
Not completed — Non-compliance with Study Drug | 0 | 0 | 4 | 1
Not completed — Pregnancy | 0 | 0 | 5 | 0
Not completed — Lack of Efficacy | 0 | 0 | 2 | 0
Not completed — HbsAg Seroconversion | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: Participants who received at least 1 dose of study drugs.
Groups:
- TAF 25 mg: Double-blind Phase: Tenofovir alafenamide (Vemlidy®; TAF) 25 mg + tenofovir disoproxil fumarate (TDF) placebo tablets administered once daily for up to 96 weeks (per amendment 1 & 2) or 144 weeks (per amendment 3).
  Open-label TAF extension Phase: After Week 96 or 144 in the Blinded Treatment Phase, participants were given the option to continue with OL TAF 25 mg for additional 288 or 240 weeks (Up to Week 384), respectively.
  After the completion of OL TAF Extension Phase treatment or when there was early discontinuation of treatment, participants either switched to commercially available anti-HBV treatments in their country or entered follow-up phase and were followed-up every 4 weeks for 24 weeks off treatment (TFFU) for the assessment of safety.
- TDF 300 mg: Double-blind Phase: TDF 300 mg + TAF placebo tablets administered once daily for up to 96 weeks (per amendment 1 & 2) or 144 weeks (per amendment 3).
  Open-label TAF extension Phase: After Week 96 or 144 in the Blinded Treatment Phase, participants were given the option to continue with OL TAF 25 mg for additional 288 or 240 weeks (Up to Week 384), respectively.
  After the completion of OL TAF Extension Phase treatment or when there was early discontinuation of treatment, participants either switched to commercially available anti-HBV treatments in their country or entered follow-up phase and were followed-up every 4 weeks for 24 weeks off treatment (TFFU) for the assessment of safety.
- Total: Total of all reporting groups
Arm/Group | TAF 25 mg | TDF 300 mg | Total
Number analyzed (Participants) | 581 | 292 | 873
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38 (11.0) | 38 (11.7) | 38 (11.3)
Age, Customized [Count of Participants; unit: Participants]
  < 50 years | 493 | 234 | 727
  >= 50 years | 88 | 58 | 146
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 210 | 103 | 313
  Male | 371 | 189 | 560
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 575 | 290 | 865
  Unknown or Not Reported | 4 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 482 | 232 | 714
  Native Hawaiian or Other Pacific Islander | 1 | 3 | 4
  Black or African American | 2 | 3 | 5
  White | 96 | 52 | 148
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Russia | 33 | 16 | 49
  Romania | 24 | 9 | 33
  Singapore | 7 | 2 | 9
  Hong Kong | 71 | 50 | 121
  United States | 33 | 21 | 54
  Japan | 35 | 11 | 46
  United Kingdom | 5 | 3 | 8
  India | 77 | 33 | 110
  Spain | 4 | 0 | 4
  New Zealand | 11 | 6 | 17
  Canada | 55 | 28 | 83
  Turkey | 15 | 11 | 26
  Taiwan | 54 | 29 | 83
  South Korea | 120 | 53 | 173
  Poland | 7 | 5 | 12
  Italy | 9 | 5 | 14
  Australia | 14 | 6 | 20
  Bulgaria | 4 | 2 | 6
  France | 3 | 2 | 5
HBV DNA [Mean (Standard Deviation); unit: log10 IU/mL] | 7.6 (1.34) | 7.6 (1.41) | 7.6 (1.36)
Plasma HBV DNA Level [Count of Participants; unit: Participants]
  < 8 log10 IU/mL | 309 | 150 | 459
  ≥ 8 log10 IU/mL | 272 | 142 | 414
IL28B Genotype [Count of Participants; unit: Participants] — The CC, CT, and TT alleles are different forms of the IL28b gene.
  Participants
    CC | 442 | 210 | 652
    CT | 112 | 69 | 181
    TT | 23 | 10 | 33
    Missing | 4 | 3 | 7
Oral Antiviral Treatment Status [Count of Participants; unit: Participants]
  Treatment Experienced | 151 | 77 | 228
  Treatment Naive | 430 | 215 | 645
Proteinuria by Urinalysis (dipstick) [Count of Participants; unit: Participants] — Urine protein was measured using the dipstick method. Grade 0 = Absent; Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe.
  Participants
    Grade 0 | 538 | 259 | 797
    Grade 1 | 40 | 31 | 71
    Grade 2 | 3 | 2 | 5
    Grade 3 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Hepatitis B Virus (HBV) DNA < 29 IU/mL at Week 48
Time Frame: Week 48
Population: Full Analysis Set: participants who were randomized into the study and received at least 1 dose of study drugs. Participants were analyzed according to the treatment to which they were randomized.
Measure: Number; unit: percentage of participants
Groups:
- TAF 25 mg: TAF 25 mg tablet + TDF placebo tablet once daily for up to 96 weeks (per amendment 1 & 2) or 144 weeks (per amendment 3).
- TDF 300 mg: TDF 300 mg tablet + TAF placebo tablet once daily for up to 96 weeks per amendment 1 & 2) or 144 weeks (per amendment 3).
Arm/Group | TAF 25 mg | TDF 300 mg
Number analyzed (Participants) | 581 | 292
percentage of participants | 63.9 | 66.8
Statistical Analysis 1: Comparison: TAF 25 mg vs TDF 300 mg; The null hypothesis was that the TAF group is at least 10% worse than the TDF group with respect to the proportion of participants with HBV DNA < 29 IU/mL at Week 48. The alternative hypothesis was that the TAF group is less than 10% worse than the TDF group with respect to the proportion of participants with HBV DNA < 29 IU/mL at Week 48. Noninferiority was assessed using a 95% confidence interval (CI) approach, with a noninferiority margin of 10%; Test type: Non-Inferiority or Equivalence — Sample sizes of 288 and 576 participants in the TDF and TAF groups, respectively, were planned to give 84% power to rule out the noninferiority margin of 10% at a 1-sided significance level of 0.025. This sample size based on the assumption that the expected difference (TAF - TDF) in the proportion of participants with HBV DNA < 29 IU/mL was 0 and the proportion of participants with HBV DNA < 29 IU/mL in the TDF group was 69%. Missing data were treated as not achieving the primary endpoint; Difference in proportions = -3.6, 95% CI 2-sided [-9.8 to 2.6] — Difference in the proportion between treatment groups and its 95% CI were calculated based on the Mantel-Haenszel (MH) proportions adjusted by baseline HBV DNA categories and oral antiviral treatment status strata

2. Secondary Outcome: Percentage of Participants With Hepatitis B e Antigen (HBeAg) Seroconversion to Antibody Against Hepatitis B e Antigen (Anti-HBe) at Week 48
Time Frame: Week 48
Population: Serologically Evaluable Full Analysis Set: participants who were randomized, had received at least 1 dose of study drug, and were HBeAg positive and anti-HBe negative or had a value missing value at baseline. Participants were analyzed according to their randomized treatment group. All missing data were treated as no HBeAg seroconversion.
Measure: Number; unit: percentage of participants
Arm/Group | TAF 25 mg | TDF 300 mg
Number analyzed (Participants) | 565 | 285
percentage of participants | 10.3 | 8.1

3. Secondary Outcome: Percent Change From Baseline in Hip Bone Mineral Density (BMD) at Week 48
Time Frame: Baseline, Week 48
Population: Participants in the Hip Dual-Energy X-ray Absorptiometry (DXA) Analysis Set (participants who were randomized, received at least 1 dose of study drugs, and had nonmissing baseline hip BMD values) with available data were analyzed. Participants were analyzed according to the treatment they actually received. Missing data were excluded from analysis.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | TAF 25 mg | TDF 300 mg
Number analyzed (Participants) | 537 | 271
percentage change | -0.100 (2.2912) | -1.715 (2.5723)

4. Secondary Outcome: Percent Change From Baseline in Spine BMD at Week 48
Time Frame: Baseline, Week 48
Population: Participants in the Spine DXA Analysis Set (participants who were randomized, received at least 1 dose of study drugs, and had nonmissing baseline spine BMD values) with available data were analyzed. Participants were analyzed according to the treatment they actually received. Missing data were excluded from analysis.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | TAF 25 mg | TDF 300 mg
Number analyzed (Participants) | 543 | 274
percentage change | -0.417 (2.9343) | -2.294 (3.1331)

5. Secondary Outcome: Change From Baseline at Week 48 in Serum Creatinine
Time Frame: Baseline, Week 48
Population: Participants in the Safety Analysis Set with available data were analyzed. Participants were analyzed according to the treatment they actually received. Missing data were excluded from analysis.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | TAF 25 mg | TDF 300 mg
Number analyzed (Participants) | 553 | 283
mg/dL | 0.009 (0.1238) | 0.026 (0.0948)

6. Other Pre Specified Outcome: Percentage of Participants With Treatment-emergent Proteinuria by Urinalysis (Dipstick) Through Week 48
Description: Grades 1 (mild), 2 (moderate), and 3 (severe) were the highest treatment-emergent postbaseline grades for urine protein using the dipstick method.
Time Frame: Up to 48 weeks
Population: Participants in the Safety Analysis Set with at least 1 postbaseline urine protein value were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | TAF 25 mg | TDF 300 mg
Number analyzed (Participants) | 577 | 286
percentage of participants
  Grade 1 | 23.9 | 17.8
  Grade 2 | 3.5 | 4.5
  Grade 3 | 0 | 0.3

ADVERSE EVENTS:
Time Frame: All-Cause Mortality: Randomization up to approximately 416 weeks; Adverse Events: First dose date up to Week 384
Description: All-cause mortality: Randomized Analysis Set: All participants randomized into the study.
  Adverse events: Safety Analysis Set: Participants who received at least 1 dose of study drug in the respective period.
Groups:
- Double-blind Phase: TAF 25 mg: TAF 25 mg + TDF placebo tablets administered once daily for up to 96 weeks (per amendment 1 & 2) or 144 weeks (per amendment 3).
- Double-blind Phase: TDF 300 mg: TDF 300 mg + TAF placebo tablets administered once daily for up to 96 weeks (per amendment 1 & 2) or 144 weeks (per amendment 3).
- Open-label TAF Extension Phase: TAF 25 mg to TAF 25 mg: After Week 96 or 144 in the Blinded Treatment Phase, participants were given the option to continue with OL TAF 25 mg for additional 288 or 240 weeks (Up to Week 384).
  After the completion of OL TAF Extension Phase treatment or when there was early discontinuation of treatment, participants either switched to commercially available anti-HBV treatments in their country or entered follow-up phase and were followed-up every 4 weeks for 24 weeks off treatment (TFFU) for the assessment of safety.
- Open-label TAF Extension Phase: TDF 300 mg to TAF 25 mg: After Week 96 or 144 in the Blinded Treatment Phase, participants were given the option to switch to Open-label (OL) TAF 25 mg for additional 288 or 240 weeks (Up to Week 384).
  After the completion of OL TAF Extension Phase treatment or when there was early discontinuation of treatment, participants either switched to commercially available anti-HBV treatments in their country or entered follow-up phase and were followed-up every 4 weeks for 24 weeks off treatment (TFFU) for the assessment of safety.
Arm/Group | Double-blind Phase: TAF 25 mg | Double-blind Phase: TDF 300 mg | Open-label TAF Extension Phase: TAF 25 mg to TAF 25 mg | Open-label TAF Extension Phase: TDF 300 mg to TAF 25 mg
All-Cause Mortality (participants affected / at risk) | 2/582 | 1/293 | 0/514 | 0/253
Serious Adverse Events (participants affected / at risk) | 44/581 | 20/292 | 59/514 | 32/253
Other Adverse Events (participants affected / at risk) | 290/581 | 143/292 | 168/514 | 100/253
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Phase: TAF 25 mg (N=581) | Double-blind Phase: TDF 300 mg (N=292) | Open-label TAF Extension Phase: TAF 25 mg to TAF 25 mg (N=514) | Open-label TAF Extension Phase: TDF 300 mg to TAF 25 mg (N=253)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 2 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 2 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Cushing's syndrome (Endocrine disorders) | 0 | 0 | 1 | 0
Goitre (Endocrine disorders) | 1 | 0 | 1 | 0
Angle closure glaucoma (Eye disorders) | 0 | 0 | 0 | 1
Macular hole (Eye disorders) | 0 | 0 | 1 | 0
Retinal detachment (Eye disorders) | 1 | 0 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Proctitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 2
Pyrexia (General disorders) | 1 | 0 | 3 | 0
Suprapubic pain (General disorders) | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 1 | 1
Hepatomegaly (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 1 | 0
Anal abscess (Infections and infestations) | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 1 | 1
Chronic sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Covid-19 (Infections and infestations) | 0 | 0 | 1 | 0
Dengue fever (Infections and infestations) | 1 | 1 | 0 | 0
Diarrhoea infectious (Infections and infestations) | 1 | 0 | 0 | 0
Echinococciasis (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Hepatitis E (Infections and infestations) | 1 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 1
Otitis externa (Infections and infestations) | 0 | 0 | 1 | 0
Pericarditis tuberculous (Infections and infestations) | 1 | 0 | 0 | 0
Periodontitis (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 3 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Scrub typhus (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0
Tuberculosis (Infections and infestations) | 0 | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Ligament injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Limb crushing injury (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 2
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Borderline mucinous tumour of ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Gastrointestinal submucosal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 2 | 3
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Ovarian fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Thymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0
Basilar artery occlusion (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebrovascular disorder (Nervous system disorders) | 0 | 0 | 1 | 0
Coma (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1 | 1 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1 | 0
Optic neuritis (Nervous system disorders) | 0 | 1 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Abortion (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Acute psychosis (Psychiatric disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 1 | 0
Stress urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1
Endometriosis (Reproductive system and breast disorders) | 2 | 1 | 0 | 0
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Pelvic adhesions (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Prostatomegaly (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Phase: TAF 25 mg (N=581) | Double-blind Phase: TDF 300 mg (N=292) | Open-label TAF Extension Phase: TAF 25 mg to TAF 25 mg (N=514) | Open-label TAF Extension Phase: TDF 300 mg to TAF 25 mg (N=253)
Diarrhoea (Gastrointestinal disorders) | 35 | 19 | 13 | 6
Dyspepsia (Gastrointestinal disorders) | 32 | 16 | 16 | 9
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 19 | 10 | 17 | 13
Nausea (Gastrointestinal disorders) | 35 | 15 | 5 | 2
Fatigue (General disorders) | 36 | 14 | 6 | 5
Nasopharyngitis (Infections and infestations) | 71 | 29 | 33 | 13
Upper respiratory tract infection (Infections and infestations) | 70 | 33 | 32 | 17
Arthralgia (Musculoskeletal and connective tissue disorders) | 39 | 22 | 24 | 15
Back pain (Musculoskeletal and connective tissue disorders) | 36 | 22 | 20 | 12
Headache (Nervous system disorders) | 59 | 30 | 32 | 20
Cough (Respiratory, thoracic and mediastinal disorders) | 48 | 24 | 15 | 19
Hypertension (Vascular disorders) | 14 | 6 | 21 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years